CLINICAL TRIAL: NCT00667875
Title: An Exploratory Study of Naltrexone Plus Aripiprazole for Alcohol Dependence
Acronym: NALAPZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Raymond F. Anton, Distringuished University Professor, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANTON-1R21AA017525-01; R21AA017525 (NIH); NIH Grant AA017525-01
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Alcoholism; Naltrexone; Aripiprazole; Substance Abuse
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Naltrexone; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator): Naltrexone
  Interventions: Drug: Naltrexone
- 3 (Active Comparator): Naltrexone + Aripiprazole
  Interventions: Drug: Naltrexone + Aripiprazole

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: 1
Drug: Naltrexone — Naltrexone (25mg or 50 mg per titration schedule)
  Arms: 2
Drug: Naltrexone + Aripiprazole — Naltrexone + Aripiprazole (5mg - 15mg per titration schedule)
  Arms: 3

SUMMARY:
The principal aim of this exploratory study is to examine whether the addition of aripiprazole to naltrexone will enhance efficacy over naltrexone alone in a 16-week randomized, placebo-controlled clinical trial, in which all subjects will be provided medical management as delivered in the COMBINE Study (Anton et al, 2006). To test whether medication treatment will reduce drinking compared to placebo treatment alone in the context of medical management and whether naltrexone plus aripiprazole will reduce drinking compared to naltrexone treatment alone in the context of medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 70
2. Subjects will meet criteria for primary alcohol dependence operationalized as follows:

   A. Meets the DSM IV criteria for alcohol dependence including loss of control over drinking (criterion 3) B. Has not had more than one previous inpatient medical detoxification
3. Consumes, on average, at least 10 standard drinks per drinking day for men and 8 drinks per day for women in the 90 days pre-screening (to select an appropriately heavy drinking population)
4. Able to maintain sobriety for four days (with or without the aid of alcohol detoxification medications) as determined by self report, collateral report, and breathalyzer measurements
5. Able to read and understand questionnaires and informed consent
6. Lives within approximately 50 miles of the study site -

Exclusion Criteria:

1. Currently meets DSM IV criteria for any other psychoactive substance dependency disorder except nicotine dependence
2. Ever abused opiates
3. Any psychoactive substance abuse, except marijuana and nicotine, within the last 30 days as evidenced by subject report, collateral report, or urine drug screen
4. Meets DSM IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder
5. Meets DSM IV current criteria for dissociative disorder or eating disorders
6. Has current suicidal ideation or homicidal ideation
7. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications
8. Current use of disulfiram
9. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problem that would impair participation or limit medication ingestion
10. Hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 3.0 times normal at screening and/or after 5 days abstinence
11. Sexually active female of child-bearing potential who is pregnant (by urine HCG), nursing, or who is not using a reliable form of birth control
12. Has current charges pending for a violent crime (not including DUI-related offenses)
13. Does not have a stable living situation and a reliable source of collateral reporting
14. Has taken an opiate antagonist drug in the last month
15. Has taken aripiprazole in the last month or has experienced adverse effects from it at any time in the past

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Center for Drug and Alcohol Programs, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the community in response to advertising in local papers, and radio
Pre-assignment Details: Subjects were to remain abstinent for 4 days prior to starting treatment with the randomly assigned study drug.
Groups:
- 1 Placebo: Placebo : placebo
- 2 Naltrexone: Naltrexone
  Naltrexone : Naltrexone (25mg or 50 mg per titration schedule)
- 3 Naltrexone Plus Aripiprazole: Naltrexone + Aripiprazole
  Naltrexone + Aripiprazole : Naltrexone + Aripiprazole (5mg - 15mg per titration schedule)
Period: Overall Study
Arm/Group | 1 Placebo | 2 Naltrexone | 3 Naltrexone Plus Aripiprazole
Started | 23 (3 subjects had no data after randomization and were excluded from analysis) | 21 | 21 (2 subjects had no data following randomization and were excluded from the analysis.)
Subjects Included in Analysisd | 20 | 21 | 19
Completed | 13 (Subjects who dropped out during treatment are considered completed if they provide end of study data) | 10 | 8
Not Completed | 10 | 11 | 13
Not completed — Adverse Event | 0 | 2 | 6
Not completed — Withdrawal by Subject | 10 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Placebo | 2 Naltrexone | 3 Naltrexone Plus Aripiprazole | Total
Number analyzed (Participants) | 23 | 21 | 21 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9.6) | 47.2 (11.3) | 48.4 (10.2) | 47.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 23
  Male | 16 | 14 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: Standard drinks per drinking day
Time Frame: 16-week treatment period
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Groups:
- Inactive Placebo: Inactive placebo naltrexone + inactive placebo Aripiprazole
- Naltrexone and Inactive Placebo Aripiprazole: Naltrexone: Naltrexone (25mg or 50 mg per titration schedule)
Arm/Group | Inactive Placebo | Naltrexone and Inactive Placebo Aripiprazole | Naltrexone + Aripiprazole
Number analyzed (Participants) | 20 | 21 | 19
drinks per drinking day | 7.2 (7.3) | 7.8 (6.6) | 5.2 (7.2)
Statistical Analysis 1: Comparison: Inactive Placebo vs Naltrexone and Inactive Placebo Aripiprazole vs Naltrexone + Aripiprazole; Analyzed as a mixed model, Group by time (4 time blocks) with an unstructured variance/covariance matrix. Baseline drinks per day was used as a covariate; Test type: Superiority; p = 0.49, Mixed Models Analysis — The p value represents variation of the total 16 week trial over all three groups

2. Primary Outcome: Percent Heavy Drinking Days
Description: percent of total 112 day trial in which heavy drinking occurred (>=4 for females, >=5 male)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percent of days
Groups:
- Placebo: Placebo: Placebo naltrexone and placebo aripiprazole
- Naltrexone: Placebo Aripiprazole: Naltrexone
  Naltrexone: Naltrexone (25mg or 50 mg per titration schedule): placebo aripiprazole
- Naltrexone:Aripiprazole: Naltrexone + Aripiprazole
  Naltrexone + Aripiprazole: Naltrexone + Aripiprazole (5mg - 15mg per titration schedule)
Arm/Group | Placebo: Placebo | Naltrexone: Placebo Aripiprazole | Naltrexone:Aripiprazole
Number analyzed (Participants) | 20 | 21 | 19
percent of days | 10.54 (20.0) | 16.7 (19.9) | 7.34 (19.7)
Statistical Analysis 1: Comparison: Placebo: Placebo vs Naltrexone: Placebo Aripiprazole vs Naltrexone:Aripiprazole; Analyzed as a mixed model (SPSS linear mixed) with an unstructured variance/covariance and baseline percent heavy drinking days as a covariate; Test type: Superiority; p = 0.03, Mixed Models Analysis — The p value represents variation of the total 16 week trial over all three groups

3. Secondary Outcome: Pill Counts During Treatment
Description: Compliance with medication as determined by pill counts
Time Frame: 16-week
Measure: Mean (Standard Deviation); unit: Percent of pills taken
Arm/Group | 1 Placebo | 2 Naltrexone | 3 Naltrexone Plus Aripiprazole
Number analyzed (Participants) | 20 | 21 | 19
Percent of pills taken
  Percent aripiprazole or aripiprazole placebo taken | 96.4 (6.5) | 97.0 (4.7) | 84.2 (25.2)
  Percent naltrexone or naltrexone placebo taken | 96.8 (5.9) | 96.9 (4.2) | 86.4 (22.7)
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Naltrexone vs 3 Naltrexone Plus Aripiprazole; Test type: Superiority — Anova across all three treatment groups; p < .05, ANOVA; Naltrexone or naltrexone placebo pills taken F=3.9 df 2 Aripiprazole or aripiprazole placebo pills taken F=4.6 df 2

4. Secondary Outcome: Percent Riboflavin Positive Urine Samples as a Measure of Medication Compliance
Description: Riboflavin was added to each individual capsule of medication and measured as a proxy for compliance with the medication regime
Time Frame: 16 weeks treatment trial
Measure: Mean (Standard Deviation); unit: Percent of riboflavin positive samples
Arm/Group | Placebo: Placebo | Naltrexone: Placebo Aripiprazole | Naltrexone:Aripiprazole
Number analyzed (Participants) | 20 | 21 | 19
Percent of riboflavin positive samples | 74.9 (33.7) | 85.1 (18.5) | 62.1 (30.9)
Statistical Analysis 1: Comparison: Placebo: Placebo vs Naltrexone: Placebo Aripiprazole vs Naltrexone:Aripiprazole; Anova across three groups; Test type: Superiority; p < .05, ANOVA; f 3.2 df 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 16 weeks following randomization visit.
Description: The SAFTEE was used to collect this data. Psychopharmacol Bull. 1986;22(2):343-81
Arm/Group | Inactive Placebo | Naltrexone and Inactive Placebo Aripiprazole | Naltrexone + Aripiprazole
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 21/23 | 20/21 | 19/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactive Placebo (N=23) | Naltrexone and Inactive Placebo Aripiprazole (N=21) | Naltrexone + Aripiprazole (N=21)
Dizziness (General disorders) | 6 (11) | 9 (17) | 10 (21)
Nausea and/or vomiting (Gastrointestinal disorders) | 6 (6) | 12 (20) | 10 (14)
Headache (General disorders) | 14 (34) | 10 (15) | 9 (20)
Fatigue or tiredness (General disorders) | 10 (37) | 16 (39) | 12 (20)
Diarrhea (Gastrointestinal disorders) | 4 (7) | 8 (15) | 3 (5)
Nervousness/anxiety (Nervous system disorders) | 12 (45) | 13 (34) | 11 (27)
Insomnia (General disorders) | 9 (40) | 12 (33) | 9 (28)
Somnolence (General disorders) | 7 (9) | 9 (17) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No